CLINICAL TRIAL: NCT04500379
Title: The Reliability and Validity of Chinese Version of FIBSER, STAR-P, HEA Scale in Depression
Brief Title: Reliability and Validity of FIBSER, STAR-P, HEA Scale The Reliability and Validity of Chinese Version of FIBSER, STAR-P, HEA Scale in Depression Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-52
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2021-09

CONDITIONS: Depression
Keywords: FIBSER; STAR-P; HEA scale
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the survey of the World Health Organization, the number of patients with depression in the world has reached 350 million, has becoming the primary cause of disability and the main disease burden worldwide. In order to better dealing with adverse reactions, improving the doctor-patient relationship and optimizing the treatment cost, FIBSER, STAR-P and HEA Health Economics Follow-up Evaluation Scale are selected as simple and quick evaluation scales to evaluate the influence, doctor-patient relationship and social and economic benefits after drug treatment in clinical treatment. At present, the reliability and validity of FIBSER, STAR-P and HEA scales will be verified the reliability and validity of the above three scales in depressive disorder, aiming at enriching the treatment of depressive patients based on assessment, thus improving the compliance of medication for depressive disorder, improving the doctor-patient relationship and reducing the total burden of social diseases.

DETAILED DESCRIPTION:
In this study, the reliability and validity of FIBSER Scale, Doctor-patient Relationship Scale-Patient Edition (STAR-P) and HEA in Chinese population will be verified to increase the diversity and selectivity of domestic assessment tools.

This study includes two steps.

1. baseline: demographic data, HAM-D, HAM-A, YMRS, drug side effects scale：FIBSER, TESS； doctor-patient relationship scale ：STAR-P, PDRQ-15；Health economics follow-up evaluation scale ：SDS and HEA were evaluated.
2. follow-up (4 weeks): HAM-D, HAM-A, YMRS, FIBSER, STAR-P and HEA scale in order to verify the reliability of retest.

ELIGIBILITY:
Inclusion Criteria:

* Case group:

  1. The subjects were psychiatric outpatients and inpatients who were able and willing to provide informed consent.
  2. Men or women aged between 18 and 65, with junior high school education or above.
  3. according to DSM-5 criteria, patients diagnosed with depressive disorder.
  4. The total score of Hamilton Depression Scale (HAM-D) was ≥7 and the total score of Young Mania Scale (YMRS) was ≤5.
  5. subjects were treated with antidepressants at least two weeks before the study visit, all of them were SSRIs.

Control group:

1）did not meet the diagnostic criteria of any axis I in DSM-5. 2）18-65 years old, with junior high school education or above. 3）Willing to participate in this study, and the subjects signed the informed consent form.

Exclusion Criteria:

- 1）severe drug allergy. 2）Suffering from some serious physical diseases adversely affects the validity of neuropsychological test data.

3）serious negative suicide concept.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depressive disorder group: The samples were from the outpatients and inpatients of Shanghai Mental Health Center and Shanghai Pudong New Area Mental Health Center from January 2020 to December 2020, and met DSM-5 diagnostic criteria. Sixty patients aged 1865 were enrolled in the group.
  Healthy control group: The sample comes from the healthy people recruited by the society who meet the entry criteria of the control group and match the gender, age and education level, and 60 cases are planned to be enrolled in the group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Symptom Scale TESS | Up to 1 week
  Common adverse drug reactions and signs were evaluated. The "severity" column was used to evaluate the severity level of symptoms from 0 to 4. The higher the severity level, the more serious the symptoms
The Frequency, Intensity, and Burden of Side Effects Rating, FIBSER | Up to 4 week
  Evaluate three areas of drug side effects through patient self-report and rank the drug impact: frequency (how many adverse reactions caused by depression drugs in the past week), intensity (how serious adverse reactions caused by depression drugs in the past week), and burden (how much adverse reactions caused by depression drugs affect your daily activities in the past week).
HEA Health Economics Follow-up Evaluation Form，HEA | Up to 4 week
  The main evaluation in the past month includes the following items: how many times have you seen a doctor (doctor), other medical personnel, whether you have been in hospital, and the number of days off due to depression and other diseases
Sheehan Disability Scale ，SDS | Up to 1 week
  Including three items, ask patients about the degree of damage caused by their current diseases/symptoms to their work, social interaction and family functions in turn; Visual simulation score of 0-10
Doctor-patient Relationship Scale-Patient Edition ，STAR-P Doctor-patient Relationship Scale-Patient Edition (STAR-P) | Up to 4 week
  The total score of STAR-P and the scores of three subscales are adopted: active collaboration (PCO: harmonious and shared understanding of goals and mutual open and trusted experiences), active clinician input (PCI: clinicians encourage, consider, support, listen and understand patients) and non-clinician input (NCI: patients can't understand clinicians), which is composed of 12 items
PDRQ-15 Scale | Up to 1 week
  There are 15 items in total, which are divided into three dimensions: patient/family satisfaction (6 items), accessibility of medical staff (7 items) and disease attitude of patients/family members.

SECONDARY OUTCOMES:
HAM-D | Up to 4 week
  To evaluate the severity of depressive symptoms by clinicians. Remission: total score < 7.
HAM-A | Up to 4 week
  To evaluate the severity of anxiety symptoms by clinicians. The total score < 6: no anxiety sympotom.
YMRS | Up to 4 week
  Assess symptoms of mania,the total score < 6: no mania sympotom.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center IRB, Shanghai, China